CLINICAL TRIAL: NCT04740866
Title: Prospective Randomized Trial of Adjuvant Radiotherapy Versus Observation After Radical Cystectomy in High Risk Urothelial Bladder Cancer
Brief Title: Adjuvant Radiotherapy Versus Observation After Radical Cystectomy in High Risk Urothelial Bladder Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed s. Zaghloul, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bladder-03
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: High-Risk Cancer; Urothelial Carcinoma Bladder
Keywords: Adjuvant Radiotherapy; Neoadjuvant chemotherapy; Radical Cystectomy; high risk Urothelial Carcinoma Bladder; Local Control; Disease Free Survival (DFS)
MeSH Terms: interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant Radiotherapy (Active Comparator): Irradiation of both the bladder tumor bed and pelvic lymph nodes using Intensity-Modulated Radiation-Therapy [IMRT] technique.
  Interventions: Radiation: Adjuvant Radiotherapy
- Observation after radical Cystectomy (No Intervention): observation following radical cystectomy

INTERVENTIONS:
Radiation: Adjuvant Radiotherapy — Irradiation of both the bladder tumor bed and pelvic lymph nodes using Intensity-Modulated Radiation-Therapy (IMRT) technique. ([50Gy in 25 fractions conventional fractionation including tumor bed & pelvic lymph nodes]
  Arms: Adjuvant Radiotherapy

SUMMARY:
This is a prospective randomized clinical trial in high risk urothelial bladder cancer to compare adjuvant radiotherapy versus observation after radical cyctectomy. This is to clarify the benefit of adjuvant radiotherapy while limiting gastrointestinal toxicities for patients with pathological high-risk bladder cancer through assessing locoregional control (LRC).

DETAILED DESCRIPTION:
This is prospective randomized trial in high risk urothelial bladder cancer that includes 2 arms. The randomization will be done by permuted block method to 2 equal comparable groups. The total number of subjects will be 50 in each arm (Total=100 subjects).

This study include patients who may receive neoadjuvant chemotherapy [Gemcitabine+Cisplatin]) or not.

Arm (1) in this study (N=50) will received irradiation of both the bladder tumor bed and pelvic lymph nodes using IMRT technique. For Arm (2) (N=50) will undergo observation following radical cystectomy.

ELIGIBILITY:
Inclusion Criteria:

Patient with muscle-invasive urothelial cancer, who received neoadjuvant chemotherapy followed by radical cystectomy and urinary diversion with negative safety margin and belongs to one or more of the categories:

* ≥ 18 years old.
* PT3 or PT4a tumors.
* Grade 3 urothelial cancer.
* Positive infiltration of the dissected pelvic lymph nodes.

Exclusion Criteria:

* Residual tumors upon cystectomy.
* Previous pelvic irradiation.
* Non-urothelial bladder tumors.
* WHO performance status above 2.
* Any psychological, familial, sociological or geographical condition that hamper compliance with the study and/ or follow up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Local Control | Two year
  2-year local-regional control rate

SECONDARY OUTCOMES:
Disease Free Survival | Two year
  2-year disease free survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Zaghloul, MD, Principal Investigator — mszagh@yahoo.com
Locations (1):
- National Cancer Institute-Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zaghloul MS, Awwad HK, Akoush HH, Omar S, Soliman O, el Attar I. Postoperative radiotherapy of carcinoma in bilharzial bladder: improved disease free survival through improving local control. Int J Radiat Oncol Biol Phys. 1992;23(3):511-7. doi: 10.1016/0360-3016(92)90005-3. PMID 1612951
- [Result] Zaghloul MS, Christodouleas JP, Smith A, Abdallah A, William H, Khaled HM, Hwang WT, Baumann BC. Adjuvant Sandwich Chemotherapy Plus Radiotherapy vs Adjuvant Chemotherapy Alone for Locally Advanced Bladder Cancer After Radical Cystectomy: A Randomized Phase 2 Trial. JAMA Surg. 2018 Jan 17;153(1):e174591. doi: 10.1001/jamasurg.2017.4591. Epub 2018 Jan 17. PMID 29188298